CLINICAL TRIAL: NCT06304168
Title: Validation of DNA Methylation Markers for the Universal and Site-Specific Guided Cancer Detection (the VANGUARD Study)
Brief Title: Validation of DNA Methylation Markers for Universal and Site-specific Guided Cancer Detection, VANGUARD Study
Status: Recruiting | Type: Observational
Sponsor: Mayo Clinic (Other)
Responsible Party: Sponsor
Other Study IDs: 19-000890; NCI-2024-00954 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); 19-000890 (Other: Mayo Clinic Institutional Review Board)
Record Dates: First submitted 2024-02-27; First posted 2024-03-12 (Actual); Last update posted 2025-09-30 (Actual); Status verified 2025-09

CONDITIONS: Hematopoietic and Lymphatic System Neoplasm; Malignant Solid Neoplasm

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- Observational: Patients undergo blood, urine, and/or residual tissue sample collection and have their medical records reviewed on study.
  Interventions: Other: Non-Interventional Study

INTERVENTIONS:
Other: Non-Interventional Study — Non-interventional study

SUMMARY:
This study explores the potential value of a new blood test approach for early detection of cancer.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. Validate candidate universal and site-specific MDMs in DNA extracted from formalin-fixed paraffin embedded primary tumor and control specimens.

II. Test MDM-based models for detection of the top 16 most lethal human cancers using a non-invasive biological medium, specifically blood.

III. Assess feasibility for detection of cancers using urine samples to assay MDMs, RNA or protein in cell free or extra-cellular vesicles; patients may be the same or unique individuals from Aim 1 and 2.

OUTLINE: This is an observational study.

Patients undergo blood, urine, and/or residual tissue sample collection and have their medical records reviewed on study.

ELIGIBILITY:
Inclusion Criteria:

* Aim 1 Tissue

  * Cases:

    * Patient has a biopsy confirmed diagnosis of target histology
    * Tissue samples from synchronous or metachronous primary cancers may be used as long as they are clearly of a different target organ.
    * Tumors from patients with an underlying genetic disorder pre-disposing to cancer may be included as long as they are stratified from those without
  * Controls:

    * Patient does not have the diagnosis of target histology
* Aim 2 Blood

  * Cases:

    * Patient has a biopsy confirmed diagnosis of target histology or radiographic criteria that are unequivocal for diagnosis (example, meets radiographic criteria for hepatocellular carcinoma)
  * Controls:

    * Patient does not have a diagnosis of the target histology
* Aim 3 Urine

  * Cases:

    * Patient has a biopsy confirmed diagnosis of target histology or radiographic criteria that are unequivocal for diagnosis (example, meets radiographic criteria for hepatocellular carcinoma)
  * Controls:

    * Patient does not have a diagnosis of the target histology

Exclusion Criteria:

* Aim 1 Tissue

  * Cases and Controls:

    * Patient has had any transplants prior to tissue collection
    * Patient has received chemotherapy class drugs within 5 years prior to tissue collection
  * Cases:

    * Patient has had radiation to the current target lesion prior to tissue collection
    * Patient has multi-centric/multi-focal breast cancer with differing genetic profiles (ER/HER2/PR status differ; if multiple masses are present and not all are tested then exclude patient)
    * Patient has bilateral breast cancer/Ductal carcinoma in situ (DCIS)
* Aim 2 Blood

  * Cases and Controls:

    * Patient has known cancer outside of the target cancer 5 years prior to blood collection (not including basal cell or squamous cell skin cancers)
    * Patient has received chemotherapy class drugs in the 5 years prior to blood collection
    * Patient has had any prior radiation therapy to the target lesion prior to blood collection
    * Patient has had a biopsy to the target organ and/or lesion within 3 days before blood collection
  * Cases:

    * Patient has had an intervention to completely remove current target pathology
    * The current target pathology is a recurrence
    * Patient has multi-centric/multi-focal breast cancer with differing genetic profiles (ER/HER2/PR status differ; if multiple masses are present and not all are tested then exclude patient)
    * Patient has bilateral breast cancer/DCIS
* Aim 3 Urine

  * Patient has known cancer outside of the target cancer 5 years prior to urine collection (not including basal cell or squamous cell skin cancers)
  * Patient has received chemotherapy class drugs in the 5 years prior to urine collection
  * Patient has had any prior radiation therapy to the target lesion prior to urine collection
  * Patient has had a biopsy to the target organ and/or lesion within 3 days before urine collection
  * The current target pathology is a recurrence
  * Patient has chronic indwelling urinary catheter
  * Patient has had a urinary tract infection within the 14 days prior to sample collection
  * If patient does not have a primary bladder, ureter or urethral cancer, patient has a history of bladder ureter, or urethral cancer
  * Cases:

    * Patient has had an intervention to completely remove current target pathology
    * The current target pathology is a recurrence
    * Patient has multi-centric/multi-focal breast cancer with differing genetic profiles [estrogen receptor (ER)/human epidermal growth factor receptor 2 (HER2)/progesterone receptor (PR)] status differ; if multiple masses are present and not all are tested then exclude patient)
    * Patient has bilateral breast cancer/DCIS

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Cancer and control patients who will be seen or treated at Mayo clinic.
Sampling Method: Non-Probability Sample
Enrollment: 6150 (Estimated)
Dates: Start 2019-05-13 (Actual); Primary Completion 2028-05-15 (Estimated); Study Completion 2028-05-15 (Estimated)

PRIMARY OUTCOMES:
Overall cancer (Y/N) - blood test | Baseline (samples collected at enrollment)
  Blood samples will be assayed for known cancer markers to explore the potential value of a new blood test approach to detecting cancer. Accuracy of results may be evaluated based on review of past, present, and future medical record information.
Overall cancer (Y/N) - urine test | Baseline (samples collected at enrollment)
  Urine samples will be assayed for known cancer markers to explore the potential value of a new urine test approach to detecting cancer. Accuracy of results may be evaluated based on review of past, present, and future medical record information.
Cancer specific site prediction - blood samples/MDM | Baseline (samples collected at enrollment)
  Blood samples will be assayed for methylated DNA markers (MDMs) to identify individual organ sites of primary tumors.
Cancer specific site prediction - urine samples/MDM | Baseline (samples collected at enrollment)
  Urine samples will be assayed for methylated DNA markers (MDMs) to identify individual organ sites of primary tumors.
Cancer specific site prediction - blood samples/RNA | Baseline (samples collected at enrollment)
  Blood samples will be assayed for ribonucleic acid (RNA) to identify individual organ sites of primary tumors.
Cancer specific site prediction - urine samples/RNA | Baseline (samples collected at enrollment)
  Urine samples will be assayed for ribonucleic acid (RNA) to identify individual organ sites of primary tumors.

CONTACTS AND LOCATIONS:
Overall Officials: John B. Kisiel, M.D., Principal Investigator — Mayo Clinic in Rochester
Locations (1):
- Mayo Clinic in Rochester, Rochester, Minnesota, United States

REFERENCES:
- See also: Mayo Clinic Clinical Trials — https://www.mayo.edu/research/clinical-trials